CLINICAL TRIAL: NCT05819567
Title: Effect of a Newly Developed Brace on Foot Biomechanics: An in Vivo Interventional Study With Dynamic Computed Tomography.
Brief Title: Effect of a Newly Developed Brace on Foot Biomechanics.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Scafoglieri Aldo, Professor, Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23086_BraceAACO
Record Dates: First submitted 2023-04-05; First posted 2023-04-19 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: Ankle Brace; Fasciitis, Plantar; Dynamic Computed Tomography; Subtalar Joint Kinematics
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Subjects (Experimental): Students and employees of the Vrije Universiteit Brussel as well as people from outside this institution will be recruited (via Flyer), contacted and asked if they will want to participate. No gender restrictions will be applied, the participants must be adult (18<age <60) and healthy.
  Inclusion Criteria:
  * Healthy volunteers;
  * 18<Age<60;
  * Exclusion Criteria:
  * Symptoms in their lower limbs in the past 6 months
  * History of foot and/or ankle conditions and/or surgery
  * Pregnancy
  Interventions: Device: Newly Developed Ankle Brace

INTERVENTIONS:
Device: Newly Developed Ankle Brace — The ankle brace is made of gripping tissue and includes two straps and one latex wedge. The purpose of this brace is to lift up the plantar arch.

SUMMARY:
For this interventional study the investigators will recruit a number of healthy volunteers with no symptoms in their lower limbs in the past 6 months and without history of foot and/or ankle conditions and/or surgery. These volunteers will undergo a single Dynamic Computerized Tomography scan session before and after the support is carried, to find out if there is a change in the kinematics of the foot. The results will be analyzed statistically.

DETAILED DESCRIPTION:
For this study the investigators will recruit 15 healthy volunteers who will be undergone a single Dynamic Computed Tomography (4DCT) scanning session before and after wearing a brace, in order to find out if there is a change in foot kinematics. Between the two scans, the subjects will wear the brace and walk for 1 minute. Data collected with the 4DCT will be processed to get 3D imaging of the Subtalar and Midtarsal Joints, needed to quantify the rotations in the three planes of the space (Cardan Angles).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers;
* 18<Age<60;
* No gender restrictions;

Exclusion Criteria:

* Symptoms in their lower limbs in the past 6 months
* History of foot and/or ankle conditions and/or surgery
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Longitudinal Arch Angle (LAA) | 1 Day
  The Longitudinal Arch Angle (LAA) is a static measurement and is the angle defined by two vectors: the first vector passing through the midpoint of the medial malleolus to the navicular tuberosity; the second passing through the midpoint of the medial aspect of the first metatarsal head to the navicular tuberosity. The value of the LAA allowed us to identify the type of foot in one of these three categories: with LAA less than 130° is considered a pronated foot posture; with a LAA between 130° and 150° is considered a typical foot structures; with LAA greater than 150° is considered a supinated foot.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Scafoglieri, Professor, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium